CLINICAL TRIAL: NCT03291041
Title: A Proof of Concept Study to Evaluate the Effects of Tasimelteon and Placebo in Travelers With Jet Lag Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-VEC-162-2102
Record Dates: First submitted 2016-09-08; First posted 2017-09-25 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Jet Lag Disorder
MeSH Terms: interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tasimelteon (Experimental): tasimelteon, administered as oral capsule(s)
  Interventions: Drug: Tasimelteon
- Placebo (Placebo Comparator): Placebo, administered as oral capsule(s)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasimelteon — capsule
  Arms: tasimelteon
Drug: Placebo — capsule
  Arms: Placebo

SUMMARY:
A Proof of Concept Study to Evaluate the Effects of Tasimelteon and Placebo in Travelers With Jet Lag Disorder

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written consent
* Men or women between 18-75 years
* Body Mass Index of ≥ 18 and ≤ 30 kg/m2

Exclusion Criteria:

* History (within the 12 months prior to screening) of psychiatric disorders
* Major surgery, trauma, illness or immobile for 3 or more days within the past month
* Pregnancy or recent pregnancy (within 6 weeks)
* A positive test for drugs of abuse at the screening visit
* Any other sound medical reason as determined by the clinical investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Vanda Investigational Site, Alameda, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Chevy Chase, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tasimelteon | Placebo
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasimelteon | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.47) | 48.2 (16.06) | 49.8 (14.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time in the First Two-Thirds of the Night on the Night(s) Most Likely to be Disrupted
Description: Measured using polysomnography (PSG) and analyzed as change from baseline. Examination of the observational phase baseline data demonstrated that Night 3 was the night most disrupted.
Time Frame: 4 days
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
minutes | 76.2 (11.213) | 41.4 (11.882)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — LS mean and p-value are from ANCOVA with treatment and time-zone-shift as main effects and baseline value as a covariate; p = 0.0354, ANCOVA; Mean Difference (Net) = 34.75

2. Secondary Outcome: Patient Global Impression of Severity (PGI-S) Day 4
Description: Self-reported global index measure analyzed as change from baseline. The baseline was the corresponding measurement in the screening flight. The PGI-S is a single question asking the subject to rate their jet-lag condition at the present time on a scale of 1 "Normal" to 4 "Severe".
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -0.71 (0.174) | -0.07 (0.183)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0168, ANCOVA; Mean Difference (Net) = -0.63

3. Secondary Outcome: Total Sleep Time in the First Two-Thirds of the Night (All 3 Nights)
Description: Measured using polysomnography (PSG) and analyzed as change from baseline. The baseline was the corresponding measurement in the screening flight.
Time Frame: 3 Days
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
Minutes | 131.4 (35.243) | 40.9 (37.774)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0785, ANCOVA; Mean Difference (Net) = 90.56

4. Secondary Outcome: Subjective Total Sleep Time on Night 3
Description: Measured using the post-sleep questionnaire on Day 4 and analyzed as change from baseline
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
Minutes | 111.9 (23.012) | 33.47 (24.555)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0225, ANCOVA; Mean Difference (Net) = 78.45

5. Secondary Outcome: Subjective Sleep Quality Night 3
Description: Measured using the post-sleep questionnaire on Day 4 and analyzed as change from baseline. Sleep quality was ranked from 1 "Poor" to 5 "Excellent" and was the subscale of the post-sleep questionnaire used to determine subjective sleep quality.
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | 1.31 (0.273) | 0.36 (0.290)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0198, ANCOVA; Mean Difference (Net) = 0.95

6. Secondary Outcome: Subjective Sleep Latency Night 3
Description: Measured using the post-sleep questionnaire on Day 4 and analyzed as change from baseline
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
Minutes | -20.6 (8.39) | 6.0 (8.76)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0347, ANCOVA; Mean Difference (Net) = -26.55

7. Secondary Outcome: Subjective Wake After Sleep Onset Night 3
Description: Measured using the post-sleep questionnaire on Day 4 and analyzed as change from baseline
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
Minutes | -81.1 (22.53) | -24.7 (24.01)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0840, ANCOVA; Mean Difference (Net) = -56.44

8. Secondary Outcome: Karolinska Sleepiness Scale Day 4
Description: Self-reported fatigue measure analyzed as change from baseline. The baseline was the corresponding measurement in the screening flight. The KSS is a single question asking the subject to rate how sleepy they feel at that moment on a 9-point scale where 1 = extremely awake and 9 = extremely sleepy/fighting to stay wake.
Time Frame: 1 Day
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -1.69 (0.388) | -0.69 (0.409)
Statistical Analysis 1: Comparison: Tasimelteon vs Placebo; Test type: Superiority; p = 0.0765, ANCOVA; Mean Difference (Net) = -1.00

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Tasimelteon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 7/13 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tasimelteon (N=13) | Placebo (N=12)
Headache (Nervous system disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03291041/Prot_SAP_000.pdf